CLINICAL TRIAL: NCT02724137
Title: A Novel Physical Therapy Administered Physical Activity Intervention After TKR: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Daniel K. White, Dr., PT, ScD, MSc, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 643239-10
Record Dates: First submitted 2016-02-23; First posted 2016-03-31 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity
Keywords: Total Knee Replacement; Physical Therapy; Fitbit®
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy Rehab and Fitbit® (Experimental): Standard outpatient physical therapy rehabilitation after total knee replacement with the addition of a Fitbit® to promote physical activity.
  Interventions: Behavioral: Fitbit®; Other: Physical Therapy Rehab
- Physical Therapy Rehab (Active Comparator): Standard outpatient physical therapy rehabilitation after total knee replacement.
  Interventions: Other: Physical Therapy Rehab

INTERVENTIONS:
Behavioral: Fitbit® — Participants can read how many steps/day they walked on the Fitbit® daily. The treating physical therapist reviews Fitbit® recorded steps from the previous week and together with the patient sets a new step goal. The physical therapist discusses barriers to meeting step goals are discussed. Self-reward for meeting step/goal is set weekly. Participants in this group will also receive 1-month phone calls for 6-months after completing physical therapy rehabilitation to discuss physical activity, set monthly step count goal, barriers to overcoming goal and to continue to develop a reward system for when the participant achieves their step count goal.
  Arms: Physical Therapy Rehab and Fitbit®
Other: Physical Therapy Rehab — Standard of care physical therapy after total knee replacement. The goals of physical therapy are to increase knee range of motion and strength, improve balance and agility, and increase daily walking. Physical therapy appointment times range from 45-60 minutes with appointments occurring 2 times a week for 6-8 weeks.

SUMMARY:
The purpose of this study is to:

1. Determine whether the Physical Therapy (PT) & Fitbit® intervention should proceed to a full-scale clinical trial. This decision will be based on three hypotheses: Treatment promise (Hypothesis 1A): People in the PT & Fitbit® will walk 1250 more steps/day and spend 7 min/day more in moderate to vigorous physical activity (MVPA) than the control at discharge and at 6 months and 12 months, Safety (Hypothesis 1B): < 5% will have adverse events because of the intervention, A research assistant will collect data on adverse events that occur from the time of randomization until the last follow-up visit 3 months after discharge from PT. An adverse event is any unfavorable or unintended diagnosis, sign, symptom, or disease temporarily associated with the study intervention, which may or may not be related to the intervention. Adverse events include any new events not present during the pre-intervention period or events that were present during the pre-intervention period which have increased in severity. Major adverse events, such as infection, re-hospitalization or development of new comorbidities will also be noted. Recruitment (Hypothesis 1C): 75 recruited, 90% to complete trial, and 85% complete visit at 6 months and 12 months.
2. To evaluate the short- and long-term adherence of the PT & Fitbit® intervention. Short-term Adherence (Hypothesis 2A): 90% of subjects in the PT& Fitbit® group will wear the Fitbit® and participate in goal setting and behavioral counseling while in PT. Long-term Adherence (Hypothesis 2B): 75% of PT & Fitbit® will wear the Fitbit® at 6 months and 12 months.
3. To quantify changes in potential underlying mechanisms for increased physical activity. (Hypothesis 3): Change in self-efficacy for physical activity, walking endurance and participation in daily activities will be associated with improvements in physical activity.
4. To assess intervention fidelity (Hypothesis 4): (4a) using the electronic medical record, the treating PT will check off that they 1) reviewed physical activity recorded by the Fitbit® and 2) discussed step goals for all study subjects randomized to the intervention group. (4b) treating PTs will be asked to audio record five-intervention interactions/week using a digital audio recorder. A research assistant will then assess whether the PT 1) reviewed physical activity and 2) discussed step goals. Lastly, the duration of the intervention will be noted.

DETAILED DESCRIPTION:
The study is a pilot study to determine the feasibility of a full trial.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 45
* Seeking outpatient physical therapy after unilateral TKR

Exclusion Criteria:

* Not interested in increasing physical activity
* Co-morbidities other than unilateral TKR that limit physical activity
* Planning on having another lower extremity surgery in the next 6 months
* Have had another lower extremity surgery in the past 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by the Actigraph GT3X monitor | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks. Also at 6-months and 12-months from discharge from physical therapy rehab.
  This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).

SECONDARY OUTCOMES:
Short term adherence to treatment as measured by physical therapist. | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks.
  This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Self report long-term adherence to treatment as measured by research assistant. | 6 months after discharge from physical therapy rehab
  This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Reporting of adverse events | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks.
  This time frame is open-ended by design. The goal is to model our trial off of current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Number participants excluded from study as measured by research assistant. | At initial physical therapy evaluation.
  Number of participants that do not meet inclusion criteria.
Reason why the participant was excluded from the study. | At initial physical therapy evaluation.
  Categories: 1) no time/too busy 2) too much trouble 3) illness (self) 4) illness family 5) not interested 6) concerned about injury/pain 7) concerned about quality of care 8) refused
Self reported kinesiophobia using the Tampa-15 Scale for Kinesiophobia. | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks.
  This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Self reported self-efficacy using the Self-Efficacy Scale for Exercise. | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks.
  This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Intervention Fidelity using electronic medical records and digital audio recordings. | During outpatient physical therapy rehab which is expected to be 8 weeks.
  The goal is to investigate how consistent the physical activity intervention is provided to the patients. Consistency will be measured using two methods. The first is to use the EMR to check if current steps/day were recorded by the treating PT. The second is to use the digital audio recording in a subset of patients to evaluate if steps/day from the past week were reviewed by the treating PT, and if a step goal was discussed for the next week. This time frame is open-ended by design. The goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).
Self reported pain catastrophizing using the Pain Catastrophizing Scale (PSC) | Initial physical therapy evaluation to discharge from outpatient physical therapy rehab which is expected to be 8 weeks.
  This time frame is open-ended by design. Our goal is to model current physical therapy practice, in which a patient after total knee replacement goes to outpatient physical therapy and receives physical therapy services based on a timeframe planned out by their treating physical therapist. Treatment is then discontinued based on the patient's clinical presentation (ie functional mobility, strength gains, range of motion gains, patient specific goals, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K White, PT, ScD, MSc, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes